CLINICAL TRIAL: NCT05303805
Title: Analgesic and Healing Effect of Topical Sevoflurane for Chronic Venous Ulcers
Brief Title: Topical Sevoflurane for Treatment of Chronic Leg Ulcers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jiri Malek, Assoc. Prof. Jiri Malek, MD, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sevoflurane in ulcers
Record Dates: First submitted 2022-02-27; First posted 2022-03-31 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Leg Ulcer
Keywords: Leg Ulcer; Sevoflurane; Pain; Healing ulcer; Microbial colonization
MeSH Terms: conditions — Leg Ulcer; Pain; Communicable Diseases | interventions — Sevoflurane

STUDY DESIGN:
Intervention Model Description: The intervention group will have sevoflurane applied at approximately 1 ml/cm2 at the start of wound treatment, the control group will only have a standard rinse solution with , with sevoflurane used to soak the absorbent material held under the distal pole of the wound to produce a typical smell of sevoflurane.
Who Masked: Participant
Masking Description: Patient will separated by a screen from the treated area. Absorbent material with sevoflurane will be held under the distal pole of the wound to produce a typical smell of sevoflurane.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical sevoflurane (Experimental): The active treatment group will have sevoflurane applied at approximately 1 ml/cm2 at the start of wound treatment,
  Interventions: Drug: Sevoflurane
- Cyteal (Active Comparator): the control group will only have a standard rinse solution with Cyteal PIERRE FABRE MEDICAMENT, France (100 ml of skin fluid contains hexamidine diisetione 100 mg, chlorohexidine digluconate (solutio 20 %) 100 mg and chlorocresol 300 mg), with sevoflurane used to soak the absorbent material held under the distal pole of the wound.
  Interventions: Combination Product: Cyteal

INTERVENTIONS:
Drug: Sevoflurane — Topical application of 1 mL sevoflurane per 1 cm2 ulcer area once or two times daily.
  Other Names: Sevorane
  Arms: Topical sevoflurane
Combination Product: Cyteal — Rinsing and cleaning of ulcer.
  Arms: Cyteal

SUMMARY:
Patients with painful non-healing leg ulcer will be enrolled in the clinical single-blinded randomized study. The active treatment group will have sevoflurane applied at approximately 1 ml/cm2 at the start of wound treatment, the control group will only have a standard rinse solution with Cyteal TM (Pierre Fabre Medicament, France). Further treatment will then be carried out in the standard manner. The duration of the study will be 5 days; if the defect heals earlier, it will be terminated early.

Exclusion criteria: allergy to sevoflurane, inability to understand the questionnaire

Parameters to be monitored will be pain intensity, microbial colonization, appearance and size of the defect

DETAILED DESCRIPTION:
A prospective single-blinded randomized study will be conducted in patients of the Dermatovenereology Clinic of the 3rd Medical Faculty of Charles University (3LF UK) and the University Hospital Kralovske Vinohrady (FNKV) with painful non-healing tibial ulcers. Pain intensity on a numerical rating scale (NRS 0-10) must be NRS>4. The envelope method will be used for randomization. To blind patients, therapy will be performed by separating patients with a drape from the treatment area of the body. As sevoflurane has a typical odor, it will only be used in the control group to soak up absorbent material held under the distal pole of the wound without skin contact. In the active treatment group, sevoflurane will be applied at the beginning of the wound treatment at approximately 1 ml/cm2 of the ulcer surface. The standard therapy used in the control group will use only Cyteal TM lavage solution, which contains hexamidine diisetione 100 mg in 100 ml, chlorhexidine digluconate 20% solution 100 mg and chlorocresol 300 mg.

The primary aim of the study will be pain relief after sevoflurane therapy. Pain intensity will be measured by NRS at 1-hour intervals (excluding sleep); decrease of 2 point for at least 4 hours will be considered significant. Secondary aim will be healing of ulcers. The effect will be controlled by elimination of pathologic microbial colonization, cleaning of the base of the wound and decreasing the size of the ulcer. Microbial colonization will be measured by microbial swab culture before application, after the 1st application before dressing and on the 5th day after application), the appearance of the defect base will be assessed by the appearance of the surface, the size of the defect will be measured in cm2.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painful (pain intensity on the numerical scale NRS 0-10 is NRS>4) non- healing tibial venous ulcers

Exclusion Criteria:

* Allergy to sevoflurane
* Inability to understand the pain-intensity questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Continuously for 5 days
  Pain intensity measured by numeric rating scale (NRS) from 0 - no pain (the best result) to 10 - the worst possible pain using a standard questionnaire

SECONDARY OUTCOMES:
Microbial colonization | Before application of treatment, after the 1st application before tibial coverage and on the 5th day after application
  Microbial smear for culture
Size of skin defect | 5 days
  Measured in cm2
Appearance of the ulcer bed | 5 days
  Epithelial tissue, granulation tissue, slough, necrotic tissue

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Málek, M.D., Principal Investigator — 3rd Medical Faculty of Charles University
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia